CLINICAL TRIAL: NCT05607030
Title: A Second Randomized Controlled Trial of Alternating Irrigation of Vancomycin Hydrochloride and Tobramycin Sulfate in Patients Undergoing Two-Stage Exchange Arthroplasty for Periprosthetic Joint Infection of the Hip or Knee
Brief Title: A Second Trial of the Abbreviated Protocol Two-Stage Exchange
Acronym: Apex-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osteal Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTX-0302
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Prosthetic-joint Infection
Keywords: Hip; Knee; Biofilm; Minimum-biofilm-eradication-concentration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to their randomization arm assignment until the completion of Stage 1 surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental (Experimental): Local antibiotic irrigation via the VT-X7 Treatment System adjuvant to two-stage exchange arthroplasty per SOC.
  Interventions: Combination Product: VT-X7 Treatment System; Procedure: Two-stage exchange arthroplasty; Drug: Experimental Antibiotics
- Control (Active Comparator): SOC for treatment of chronic PJI - two-stage exchange arthroplasty: surgical removal of the infected implant, aggressive debridement, and exchange arthroplasty with administration of adjuvant systemic antibiotics and temporary antibiotic-impregnated cement spacer.
  Interventions: Procedure: Two-stage exchange arthroplasty; Drug: SOC Antibiotics

INTERVENTIONS:
Combination Product: VT-X7 Treatment System — Seven-day local antibiotic irrigation (alternating vancomycin hydrochloride and tobramycin sulfate) via the temporary VT-X7 Knee or Hip Spacer.
  Arms: Experimental
Procedure: Two-stage exchange arthroplasty — Stage 1 consists of surgical removal of the infected prosthesis, debridement, and implantation of a temporary spacer. Stage 2 surgery consists of explantation of the temporary spacer, debridement, and implantation of a permanent prosthesis.
Drug: SOC Antibiotics — Administration of at least 6 weeks of systemic antibiotics post-Stage 1 surgery followed by a 2-week antibiotic holiday before the Stage 2 surgery. After Stage 2 surgery, administration of at least 12 weeks of systemic antibiotics. Antibiotics will be selected by the treatment provider based on the infecting organism and administered per national and local treatment guidelines.
  Arms: Control
Drug: Experimental Antibiotics — After Stage 2 surgery, administration of at least 12 weeks of systemic antibiotics. Antibiotics will be selected by the treatment provider based on the infecting organism and administered per national and local treatment guidelines.
  Arms: Experimental

SUMMARY:
Apex-2 is a multi-site, parallel group, randomized trial. Patients will be randomly assigned in a 1:1 ratio to the Experimental Arm or the Control Arm.

The objective of the study is to evaluate safety and determine efficacy of the VT-X7 system. Efficacy is evaluated as superiority of the Experimental Arm in a composite endpoint of Overall Success at 180 days, consisting of a revision prosthesis implanted at Stage 2, absence of periprosthetic joint infection (PJI), absence of continued antibiotic therapy for treatment or prophylaxis of PJI, absence of revision surgery and absence of mortality. Secondary objectives are to evaluate overall success at 365 days, overall safety of the VT-X7 procedure, quality of life (QoL), and patient survival. The exploratory objective is to compare Experimental and Control Arms in exploratory endpoints.

Follow-up: Patients will be evaluated at 90-, 180-, and 365-day follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for two-stage exchange arthroplasty due to hip or knee periprosthetic joint infection (PJI)
* Signed informed consent
* 22 to 84 years of age (inclusive)
* Medical clearance for surgery
* Preoperative diagnosis of PJI of the hip or knee per the International Consensus Meeting of Musculoskeletal Infection (ICMMI) 2018 definition of Periprosthetic Hip and Knee Infection

Exclusion Criteria:

* Patients with 2 or more prior exchange arthroplasties (septic or aseptic) of the infected joint. Exchange of modular components only is not considered an exchange arthroplasty;
* Patients with 2 or more prior failed spacers for PJI;
* Patients for whom a Stage 2 procedure within one year is contraindicated;
* Patients with a medical history or current medical condition that requires a planned prescription of suppressive antibiotics to treat PJI of the index joint for > 12 months post Stage-2 surgery;
* Patients with bacteremia or positive bacterial blood culture in the last 30 days;
* Patients with concurrent PJI of more than one joint;
* Patients with ongoing active infection of an intravenous (IV) site;
* Patients who require long-term anticoagulation or antiplatelet therapy, and for whom bridging or withholding therapy is not recommended based on the individual's clinical condition;
* Patients with advanced renal insufficiency (i.e., chronic kidney disease Stage 4 or 5 or patients with an estimated glomerular filtration rate <30 mL/min);
* Patients on chemotherapy for malignant disease;
* Patients on systemic glucocorticoid therapy (prednisone >10 mg/day or equivalent);
* Patients who are immunodeficient (e.g., splenectomy, sickle cell anemia, Stage 3 human immunodeficiency virus infection, primary immunodeficiency disease), except patients who are immunodeficient due to immunosuppressive therapy;
* Patients who have an allergy to vancomycin hydrochloride or tobramycin sulfate (Note: prior history of red man syndrome is not considered an allergy);
* Patients who have an allergy to titanium, titanium alloys, polymethylmethacrylate or polyurethane;
* Patients who are pregnant or planning to become pregnant in the next 12 months;
* Patients with a fungal PJI as determined by one or more positive fluid and/or tissue cultures;
* Patients who have a skeletal defect greater than 150 mm in length in the tibia or femur of the infected joint;
* Patients who have a planned surgical procedure within 6 months of enrollment that can impact the conduct of the study;
* Patients who are breastfeeding;
* Patients who are incarcerated or are facing impending incarceration;
* Patients who have been in treatment or referred to treatment for substance abuse within the past year;
* Patients with any medical condition, including schizophrenia or another psychiatric disorder with hallucinations and/or delusions, that would interfere with the interpretation of the study results, the conduct of the study, or patient participation would not be in the best interest of the patient in the opinion of the Study Site Principal Investigator;
* Patients who will participate in another clinical study of an investigational drug or investigational device or have participated in another clinical study of an investigational drug or investigational device within the past 30 days that would interfere with the interpretation of the study results or the conduct of the study;
* Patients who are judged by the Study Site PI to be unsuitable for the study;
* Patients receiving immunosuppressive drug therapy for bone marrow or another transplant;
* Patients currently or previously enrolled in this study or the APEX study (JPS-0301);
* Patients who receive therapy including any of the following biologic agents, which will not be withheld for a period beginning at least one dosing cycle (minimum 7 days) prior to planned surgery and ending at least 14 days following planned surgery:

Adalimumab (Humira); Tocilizumab (Actemra); Etanercept (Enbrel); Anakinra (Kineret); Golimumab (Simponi); Secukinumab (Cosentyx); Infliximab (Remicade); Ustekinumab (Stelara); Abatacept (Orencia); Rituximab (Rituxan); Certolizumab (Cimzia); Tofacitinib (Xeljanz); Belimumab (Benlysta)

Ages: 22 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Overall Treatment Success | 180 days
  * Stage 2 revision prosthesis implanted and
  * Absence of PJI post-Stage 2 and
  * Absence of continued antibiotic therapy for treatment or prophylaxis of PJI and
  * Absence of revision surgery of the affected joint pre- and post-Stage 2 and
  * Absence of mortality.

SECONDARY OUTCOMES:
Overall Treatment Success | 365 days
  * Stage 2 revision prosthesis implanted and
  * Absence of PJI post-Stage 2 and
  * Absence of continued antibiotic therapy for treatment or prophylaxis of PJI and
  * Absence of revision surgery of the affected joint pre- and post-Stage 2 and
  * Absence of mortality.
Adverse Event Rate | 365 days
  Comparison of the cumulative proportion of subjects with reported adverse events between the study arms.
Quality Adjusted Life Years | 365 days
  Comparison of Quality Adjusted Life Years between the study arms as estimated by EQ-5D-3L.
Survival | 365 days
  Comparison of the survival between the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Piuzzi, MD, Principal Investigator — The Cleveland Clinic
Locations (19):
- United States (19):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Harbor UCLA Medical Center, Los Angeles, California
  - Kennedy White Orthopaedic Center, Sarasota, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Covenant Medical Center, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - NYU Langone Health, New York, New York
  - OrthoCarolina, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital - TriHealth Hatton Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - INTEGRIS Health Southwest Medical Center, Oklahoma City, Oklahoma
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Medical Center, Houston, Texas
  - University of Virginia Health, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No